CLINICAL TRIAL: NCT00716989
Title: LBP003: Characteristics of the Changes in the Cutaneous Immune System After Intradermal Antigen Injections
Brief Title: Pathophysiological Study of Characteristics of the Changes in the Cutaneous Immune System After Intradermal Antigen Injections
Acronym: LBP003
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Third group realisation has not been necessary regarding the results of the first two groups (no sufficient modifications in the immune response)
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Jean-François NICOLAS, MD, Hospices Civils de Lyon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2006.457
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Healthy; Immunosuppressed
Keywords: Cutaneous immune system; innate immunity; tuberculin skin tests; intradermal vaccination; pathophysiology; Healthy subjects; Immunosuppressed patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Tuberculin antigen — 2 intradermal injection of 50µl of antigen + 2 intradermal injection of 50µl of physiological serum

SUMMARY:
The goal of the vaccination is to induce humoral (antibody) and intracellular (T lymphocyte) responses. Various data show that intradermal vaccination is more efficient than intramuscular vaccination: the humoral response is statistically better after intradermic vaccination, compared to intramuscular vaccination, even in target populations such as older subjects or immunosuppressed patients

DETAILED DESCRIPTION:
Realisation of 2 groups of healthy subjects with 2 intradermal injection of 50 µl of tuberculin + 2 intradermal injection of 50 µl of physiological serum. 5 biopsy performed on 2 Tuberculin injection site, 2 physiological serum site and 1 on healthy skin site :

* Group A : healthy young subjects(18 to 40 years old) : 18 subjects
* Sub-group A1 (biopsy 30 minutes after injection) : 6 subjects
* Sub-group A2 (biopsy 4 hours after injection) : 6 subjects
* Sub-group A3 (biopsy 72 hours after injection) : 6 subjects
* Group B : healthy old subjects(60 to 75 years old) : 18 subjects
* Sub-group B1 (biopsy 30 minutes after injection) : 6 subjects
* Sub-group B2 (biopsy 4 hours after injection) : 6 subjects
* Sub-group B3 (biopsy 72 hours after injection) : 6 subjects

Determination of the best time (30 minutes, 4 hours or 72 hours)for intradermal vaccination caracteristics after group A and B data analysis. From these results, last group of immunosuppressed patients performed:Group C with 6 immunosuppressed patients (18 to 60 years old)

ELIGIBILITY:
Inclusion Criteria:

* Both genders eligible for study.
* Female participants must use a contraceptive method.
* Tuberculin skin test between 1 and 15mm
* Participants must be able to understand and sign the Informed Consent, and comply with all aspects of the protocol.
* Subjects registered in a social security system or with health insurance cover
* First group: Healthy subjects aged from 18 to 75 years with 2 subgroups: 18-40 and 60-75 year old subjects
* Second group: Patients with kidney transplants of longer than 6 months on immunosuppressive treatment

Exclusion Criteria:

* Pregnant or lactating women.
* Previous allergic reaction to tuberculin skin test
* Active skin disease on testing zone
* Patients with a clinically significant disease (chronic, recurrent or active)
* Local or systemic medication which interacts with the outcome measures.
* Patients deprived of their civic rights, in custody, or under the care of a tutorial, judiciary or administrative body.
* Patients relevant of a protection measure
* Patients in a critical medical situation
* Patients with a personal situation evaluated by the investigator as unable to give an optimal participation in the study, or where it could constitute a risk for the patient
* Linguistic barrier or psychological profile disabling the patient from signing the consent form
* Patient still in an exclusion period following participation in another clinical trial
* Patients having earned more than 4500€ in indemnities following participation in clinical trials during the last 12 months, including this study

For group 1 only:

* Systemic corticotherapy or immunosuppressive treatment within the 2 weeks before first visit or within 2 weeks before the third visit or the biopsies.
* Systemic non anti-inflammatory drugs the week before the first visit or within 1 week before the third visit or the biopsies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Cellular changes of recruited cells by immunochemical and histological analysis in the three groups of subjects (healthy young subjects, healthy old subjects and immunosuppressed patients) | 30 minutes, 4 hours or 72 hours

SECONDARY OUTCOMES:
Molecular analysis of cytokines and chemokines involved in recruitment and/or function of immunocompetent cells | 30 minutes, 4 hours or 72 hours
Comparison of changes in the cutaneous immune system between the three groups of subjects | 30 minutes, 4 hours or 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François NICOLAS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France